CLINICAL TRIAL: NCT05180500
Title: Phase 1 Clinical Trial of a Q GRFT Nasal Spray
Brief Title: Safety and Acceptability of Q GRFT Nasal Spray for COVID-19 Prophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sharon Hillier (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Hillier, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY21100009; 3P30CA047904-32S5 (NIH)
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Pharmacokinetics; Safety
Keywords: Intranasal spray; Prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — q-griffithsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Q-GRFT Nasal Spray (Active Comparator): Q-Griffithsin (Q-GRFT) nasal spray (7.5mg/mL). Two metered doses of 100μL into each nostril, total of 3mg Q-GRFT per administration, administered once daily for 14 consecutive days.
  Interventions: Drug: Q-Griffithsin
- Placebo Nasal Spray (Placebo Comparator): Placebo Nasal Spray. Two metered doses of 100μL into each nostril, administered once daily for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q-Griffithsin — Q-Griffithsin is derived from Griffithsin (GRFT) which is a non-glycosylated protein consisting of 121 amino acids. Q-GRFT contains a single amino acid substitution, M78Q variant, resistant to oxidation yet maintains the parent molecule's pharmacological profile.
  Arms: Q-GRFT Nasal Spray
Drug: Placebo — A matched vehicle solution manufactured and dispensed in same applicators as the active comparator.
  Arms: Placebo Nasal Spray

SUMMARY:
This is a phase I randomized, placebo-controlled, single site to assess the local and systemic safety of intranasal Q-Griffithsin (Q-GRFT) after 14 doses in approximately 45 adult participants. Participants will be randomized 2:1 (Q-GRFT nasal spray: placebo nasal spray) resulting in 30 participants enrolled into the Q-GRFT arm and 15 participants enrolled into the placebo arm. A clinician will apply two metered doses of Q-GRFT in each nostril (400μl total) of the participant on the day of enrollment. Participants will be monitored in the clinic for 1 hour after administration and return for a 24-hour post dose visit. If safe and acceptable, a second period of daily administration by the participant for 13 days will commence. Safety assessments will be performed at day 7, day 14, and day 28 visits after the initiation of the second period. The expected duration of study participation for each participant will be approximately 6-8 weeks. The primary endpoint is the proportion of participants who experience a related Grade 2 or higher adverse event. Secondary and exploratory endpoints include persistence and systemic absorption of Q-GRFT, acceptability and the impact of Q-GRFT nasal spray on smell.

DETAILED DESCRIPTION:
This is a phase 1 study for intranasal application of Q-Griffithsin (Q-GRFT) spray as a prophylactic for severe acute respiratory syndrome-CoV-2. This randomized, placebo-controlled, single site will assess the local and systemic safety of intranasal Q-GRFT after 14 doses in approximately 45 adult participants. Participants will be randomized 2:1 (Q-GRFT nasal spray: placebo nasal spray) resulting in 30 participants enrolled into the Q-GRFT arm and 15 participants enrolled into the placebo arm. Accrual of approximately 45 evaluable participants is expected to take 6 months. The expected duration of study participation for each participant will be approximately 6-8 weeks. A clinician will apply two metered doses of Q-GRFT in each nostril (400μl total) of the participant on the day of enrollment. Participants will be monitored in the clinic for 1 hour after administration and return for a 24-hour post dose visit. If safe and acceptable, a second period of daily administration by the participant for 13 days will commence after a 5-49 day washout period. Safety assessments will be performed at day 7, day 14, and day 28 visits after the initiation of the second period. Additional safety assessments will be done by contacting participants between the 24-hour and 7-day visits and 7- and 14-day visits. The expected duration of study participation for each participant will be approximately 6-8 weeks. The primary endpoint is the proportion of participants who experience a related Grade 2 or higher adverse event. Secondary and exploratory endpoints include persistence and systemic absorption of Q-GRFT, acceptability and the impact of Q-GRFT nasal spray on smell.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* In general good health as determined by the site clinician
* Negative SARS-CoV-2 test at screening
* Fully vaccinated for SARS-CoV-2 (does not include booster vaccination)
* Agree to abstain from any other investigational drug studies for the duration of the study
* Agree to abstain from nasally administered products, including over-the-counter products, for the duration of the study
* Report use of an effective method of contraception at enrollment and intending to continue use of an effective method for the duration of study participation. Acceptable methods include:

  1. Males: Male condoms, sterilization of participant or partner, partner use of hormonal contraception or intrauterine device, identifies as a man who has sex with men exclusively, and/or sexually abstinent for the past 60 days and agrees to remain abstinent for the study duration
  2. Females: Hormonal methods at the time of enrollment, intrauterine device inserted prior to enrollment, sterilization of participant or partner, consistent condom use of male partner for at least 28 days (reports using condoms 10 times in the last 10 acts of intercourse), identifies as a woman who has sex with women exclusively, and/or sexually abstinent for the past 60 days and agrees to remain abstinent for the study duration.
* Agree to participate in all study-related assessments and procedures

Exclusion Criteria:

* Abnormal nasal or throat exam at enrollment
* If female, pregnancy, or within 42 days of last pregnancy at screening
* If female, breastfeeding
* Diagnosed with SARS-CoV-2 in the past 42 days at screening
* Diagnosed or suspected respiratory tract infection in the past 14 days at screening (including asymptomatic SARS-CoV-2)
* Participation in an investigational drug study in past 30 days at screening
* Any condition that, in the opinion of the Investigator would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
* Use of any intranasal product in the 14 days prior to enrollment
* Surgical procedure involving the nose or throat 90 days prior to enrollment
* Any of the following laboratory abnormalities at screening:

  1. Hgb < 12g/dL (men) and < 11g/dL (women)
  2. Serum creatinine > 1.1 x upper limit of normal
  3. alanine transaminase, aspartate aminotransferase, and total bilirubin > 1.1 x upper limit of normal
* Grade 2 or higher seasonal allergies at the time of enrollment
* Reported use of illicit drugs

  1. Non-therapeutic injection drug use in the 12 months prior to screening
  2. Any use of methamphetamine, gamma hydroxybutyrate, cocaine or heroin in the 12 months prior to screening
* Use of systemic prescription immunomodulatory medications within the 4 weeks prior to the enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Ingrid Macio, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Started | 33 | 17
Completed | 30 | 17
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 33 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 32 | 17 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (7.7) | 27.6 (6.3) | 28.1 (7.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity by participant report
  Participants
    Female | 23 | 11 | 34
    Male | 10 | 4 | 14
    Nonbinary | 0 | 1 | 1
    Transgender male to female | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 23 | 12 | 35
    Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 32 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 21 | 12 | 33
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 17 | 50
COVID-19 Diagnosis [Count of Participants; unit: Participants] — Participant received one or more positive diagnoses for COVID-19 in the past
  Participants
    Yes | 11 | 6 | 17
    No | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Related Grade 2 or Higher Adverse Events
Description: Number of participants with Grade 2 or higher adverse events deemed related to study product
Time Frame: Approximately 8 weeks
Population: All participants randomized to study product are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 33 | 17
Participants
  Participants with related Grade 2 or higher | 6 | 2
  Participants without related Grade 2 or higher | 27 | 15
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = .70, Fisher Exact

2. Secondary Outcome: Q-GRFT Concentration From Nasopharyngeal Swab Eluent Collected at 24 Hours
Description: Q-GRFT concentration from nasopharyngeal swab eluent collected 24 hours after intranasal application of a single dose of study product.
Time Frame: Approximately 24 hours
Population: All participants on whom a nasopharyngeal swab was collected 24 hours after intranasal application of a single dose of study product.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 31 | 17
ng/mL | 1007 [NA to 1740] — Q-GRFT levels in 12 of 31 (39%) nasopharyngeal samples were below the limit of quantitation for the assay which was 15 ng/mL | NA [NA to NA] — Q-GRFT levels in all nasopharyngeal samples were below the limit of quantitation for the assay which was 15 ng/mL
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Concentrations that were below the lower limit of quantification (<15 ng/mL) were set to 7.5 ng/mL for analyses; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Q-GRFT Plasma Concentration Collected at 24 Hours After 13 Consecutive Daily Intranasal Applications
Description: Q-GRFT concentration in plasma collected 24 hours after the final intranasal application of 13 consecutive once daily administrations of study product.
Time Frame: 24 hours after final dose of study product
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
ng/mL | NA [NA to NA] — Q-GRFT levels in all plasma samples were below the limit of quantitation for the assay which was 3ng/mL | NA [NA to NA] — Q-GRFT levels in all plasma samples were below the limit of quantitation for the assay which was 3ng/mL

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve of Q-GRFT
Description: Area under the plasma concentration versus time curve of Q-GRFT collected after 13 consecutive daily intranasal applications of study product. Q-GRFT concentrations will be measured prior to the first application of study product and at 7-days, 14-days, and 28-days after the first of thirteen daily applications of study product.
Time Frame: Approximately 28 days
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Median (Inter-Quartile Range); unit: ng x day/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
ng x day/mL | NA [NA to NA] — Q-GRFT levels in all plasma samples at all time points were below the limit of quantitation for the assay which was 3ng/mL | NA [NA to NA] — Q-GRFT levels in all plasma samples at all time points were below the limit of quantitation for the assay which was 3ng/mL

5. Secondary Outcome: Acceptability of the Intranasal Spray
Description: The acceptability of the nasal spray for use at home by the participant if it could protect against infection from coronavirus/COVID-19 will be assessed on a 5-point Likert scale, with 1 being completely unacceptable and 5 being highly acceptable. Acceptability will be assessed approximately 24 hours after the final application of 13 consecutive daily applications of the study product.
Time Frame: Approximately 14 days
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
Participants
  Acceptable (Highly or somewhat) | 26 | 17
  Unacceptable (Completely, somewhat, or neutral) | 4 | 0
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.28, Fisher Exact

6. Other Pre Specified Outcome: Mean Change in Brief Smell Identification Test (BSIT) Score
Description: Mean change in Brief Smell Identification Test (BSIT) score between the score measured before the first application of study product and measured after 13 consecutive daily applications. The BSIT score is the number of odors that a participant correctly recognizes, ranging from 0 to 12. A negative value in the change score indicates a decrease in BSIT score from the pre-dose measurement, while a positive value indicates an increase in BSIT score.
Time Frame: Approximately 14 days
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
score on a scale | -0.40 (1.10) | -0.24 (0.83)
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.60, t-test, 2 sided

7. Other Pre Specified Outcome: Q-GRFT Concentration From Nares Swab Eluent Collected at 24 Hours
Description: Q-GRFT concentration from nares swab eluent collected 24 hours after intranasal application of a single dose of study product.
Time Frame: Approximately 24 hours
Population: All participants on whom a nares swab was collected 24 hours after intranasal application of a single dose of study product.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 31 | 17
ng/mL | 1488 [NA to 6333] — Q-GRFT levels in 12 of 31 (39%) nares samples were below the limit of quantitation for the assay which was 15 ng/mL | NA [NA to NA] — Q-GRFT levels in all nares samples were below the limit of quantitation for the assay which was 15 ng/mL
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Concentrations that were below the lower limit of quantification (<15 ng/mL) were set to 7.5 ng/mL for analyses; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Q-GRFT Concentration From Nasopharyngeal Swab Eluent Collected at 24 Hours After 13 Consecutive Daily Intranasal Applications
Description: Q-GRFT concentration from nasopharyngeal swab eluent collected 24 hours after the last dose of 13 consecutive daily intranasal applications of study product.
Time Frame: Approximately 14 days
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
ng/mL | 974 [NA to 2096] — Q-GRFT levels in 8 of 30 (27%) nasopharyngeal samples were below the limit of quantitation for the assay which was 15 ng/mL | NA [NA to NA] — Q-GRFT levels in all nasopharyngeal samples were below the limit of quantitation for the assay which was 15 ng/mL
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Concentrations that were below the lower limit of quantification (<15 ng/mL) were set to 7.5 ng/mL for analyses; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Q-GRFT Concentration From Nares Swab Eluent Collected at 24 Hours After 13 Consecutive Daily Intranasal Applications
Description: Q-GRFT concentration from nares swab eluent collected 24 hours after the last dose of 13 consecutive daily intranasal applications of study product.
Time Frame: Approximately 14 days
Population: The 3 participants in the Q-GRFT arm that withdrew from the study were excluded.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 30 | 17
ng/mL | 1586 [NA to 3214] — Q-GRFT levels in 10 of 30 (33%) nares samples were below the limit of quantitation for the assay which was 15 ng/mL | NA [NA to NA] — Q-GRFT levels in all nares samples were below the limit of quantitation for the assay which was 15 ng/mL
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Concentrations that were below the lower limit of quantification (<15 ng/mL) were set to 7.5 ng/mL for analyses; Test type: Other; p < .001, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: Q-GRFT Concentration From Rectal Swab Eluent Collected at 24 Hours After 13 Consecutive Daily Intranasal Applications
Description: Q-GRFT concentration from rectal swab eluent collected 24 hours after the last dose of 13 consecutive daily intranasal applications of study product.
Time Frame: Approximately 14 days
Population: Twenty out of 50 participants consented to provide a rectal swab sample.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 6
ng/mL | 106.7 [18.3 to 510.2] | 3.4 [3.0 to 3.8]
Statistical Analysis 1: Comparison: Q-GRFT Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks.
Arm/Group | Q-GRFT Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/17
Other Adverse Events (participants affected / at risk) | 29/33 | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q-GRFT Nasal Spray (N=33) | Placebo Nasal Spray (N=17)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 22 (29) | 6 (7)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 8 (8)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (7)
Increased Sneezing (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Edematous Nasal Turbinates (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Blood on Nasopharyngeal Swab (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05180500/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT05180500/ICF_001.pdf